CLINICAL TRIAL: NCT03886415
Title: A Phase 2,Multi-center, Open-label Study Evaluating Safety and Efficacy of Jaktinib Hydrochloride Tablets in Intermediate-risk and High-risk Myelofibrosis.
Brief Title: Jaktinib Hydrochloride Tablets in Intermediate-risk and High-risk Myelofibrosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK002
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaktinib hydrochloride tablets 1 (Experimental): This is the dose group was given once a day. Jaktinib hydrochloride tablets 1 200mg qd dose group
  Interventions: Drug: Jaktinib hydrochloride tablets
- Jaktinib hydrochloride tablets 2 (Experimental): This is the dose group was given twice a day. Jaktinib hydrochloride tablets 2 100mg bid dose group
  Interventions: Drug: Jaktinib hydrochloride tablets

INTERVENTIONS:
Drug: Jaktinib hydrochloride tablets — Jaktinib hydrochloride tablets 100mg bid dose group and Jaktinib hydrochloride tablets 200mg qd dose group

SUMMARY:
This was an open-label, multi-center, randomized phase 2 study. This is a two-stage design.In the first stage, two dose groups were set up, the 100 mg bid dose group and the 200 mg qd dose group, which were randomized at 1:1, with 50 subjects in each group, and a total of 100 cases in the two groups. In the second stage, approximately 36 subjects were added to the randomized group.

DETAILED DESCRIPTION:
According to the results of the interim analysis of the ZGJAK002 of Jaktinib, a comprehensive evaluation of the benefits and risks of subjects in the 100mg bid and 200mg qd groups, the investigator and the sponsor decided to expand the enrollment of approximately 36 subjects taking 100mg bid.

ELIGIBILITY:
Inclusion criteria:

1、18 years age or older ,male or female;

2、Patients diagnosed with Primary Myelofibrosis according to WHO standard (2016 version), or patients diagnosed with Post-Polycythemia Vera Myelofibrosis or Post-Essential Thrombocythemia Myelofibrosis according to International Working Group Myeloproliferative Neoplasms Research and Treatment(IWG-MRT) standard. Both Janus Kinase 2(JAK2)mutation and JAK2 wild can be enrolled；

3、According to Dynamic International Prognostic Scoring System plus(DIPSS-plus) risk grouping criteria, patients with medium-risk-2 or high-risk myelofibrosis were assessed,Patients with grade 1 medium-risk myelofibrosis with hepatosplenomegaly and no response to existing treatment and requiring treatment can also be enrolled;

4、Subjects did not have a recent stem cell transplant program;

5、a life expectancy > 24 weeks;

6、Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2；

7、Splenomegaly: palpation of the splenic margin to or above the subcostal at least 5 cm；

8、Peripheral blood protocells ≤10%；

9、Patients who have not previously been treated with JAK inhibitors；

10、Absolute neutrophil count（ANC） ≥1000/uL, platelet count ≥75 × 109/L without growth factor, platelet production factor or platelet infusion.Subjects did not receive growth factor infusion within 2 weeks before randomization;

11、Seven days before randomization, the main organs were functioning normally, which met the following criteria： alanine transaminase（ALT）and aspartate aminotransferase（AST）≤2.5×upper limit of normal (ULN)； direct bilirubin（DBIL）and total bilirubin (TBIL)≤1.5×upper limit of normal (ULN）；serum creatinine ≤2.5×upper limit of normal (ULN)，calculated creatinine clearance（CrCl）≥50mL/min；

12、 Voluntarily sign informed consent in accordance with the requirements of the ethics committee;

13、Ability to follow study and follow-up procedures；

Exclusion Criteria:

1. Any significant clinical or laboratory abnormalities that the investigator considers to affect safety assessment, such as: a. uncontrolled diabetes (> 250 mg/dL, or 13.9 mmol > / L), b. had high blood pressure and antihypertensive drug treatment under two or unable to descend to the ranges (systolic blood pressure < 160 mmHg, diastolic pressure < 100 mmHg), c. peripheral neuropathy (NCI - CTC AE v4.03 standard grade 2 or above), d. thyroid dysfunction (> NCI - CTC AE v4.03 standard grade 2 or above);
2. The patients had a history of congestive heart failure, uncontrollable or unstable angina or myocardial infarction, cerebrovascular accident or pulmonary embolism in the first 6 months;
3. Screening of patients who have not fully recovered from surgery within the first 4 weeks;
4. Screening for patients with arrhythmia requiring treatment or QTc interval (QTcB) >480ms;
5. Screening for bacterial, viral, parasitic or fungal infections with any clinical symptoms that require treatment;
6. Patients with a history of congenital or acquired hemorrhagic diseases;
7. Patients who had previously undergone splenectomy or who had received radiotherapy of the splenic region within the first 12 months of screening;
8. Screening for HIV positive, active hepatitis b virus positive (HBsAg positive, hbv- dna positive or greater than 1000 copies /ml), anti-hcv antibody or hcv-rna positive;
9. Patients suffering from epilepsy or using psychotropic or sedative drugs at the time of screening;
10. Women who are planning to become pregnant or who are pregnant or breast- feeding, as well as those who were unable to use effective contraceptives throughout the trial;Male patients who do not use condoms during the administration and within 2 days (approximately 5 half-lives) after the last administration;
11. Patients who have suffered from malignant tumors (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) in the past 5 years;
12. Combined with other serious diseases, the researchers believe that patients' safety or compliance may be affected;
13. Suspected allergic to Jakatinib hydrochloride or similar drugs;
14. Patients who have participated in the clinical trials of other new drugs or medical devices within the first 3 months;
15. Patients who were treated with any MF drug (e.g., hydroxyl urea), any immunomulator (e.g., thalidomide), any immunosuppressant, prednisone at or above 10mg/ day or equivalent bioactive level of glucocorticoid, growth factor (e.g.,erythropoietin ), or who were within 6 half-lives of the drug within 2 weeks prior to randomization;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
effective rate | 24 weeks
  The proportion of all subjects whose spleen volume decreased by 35% or more at 24 weeks

SECONDARY OUTCOMES:
Overall response rate （CR+PR） | 24 weeks
  IWG-MRT efficacy criteria
The spleen response | 24 weeks
  The time from baseline to the first splenic volume reduction was greater than or equal to 35%；Optimal response: the proportion of patients whose spleen volume decreased by more than 35% compared with the baseline at least once;Effective time: the time from the randomization date to the first time the spleen volume decreased by more than 35% from the baseline；DoMSR: the time between the first occurrence of spleen volume reduction of more than 35% from the baseline to the increase of spleen volume less than 35% from the baseline;
Anemia response | 24 weeks
  Baseline proportion of patients with blood transfusion dependence converted to patients without blood transfusion dependence（Patients without blood transfusion dependence: patients without red blood cell transfusion for more than 12 weeks during the treatment period and with HGB ≥85g/L）;The proportion of patients with baseline non-transfusion dependence (HGB ≤100g/L) whose HGB increased by 20g/L;RBC Infusion dependence decreased: RBC infusion frequency decreased by 50%;
MF related symptom response rate | 24 weeks
  MPN-SAF TSS the proportion of patients whose total symptom score of the scale decreased by more than 50%;MPN-SAF TSS the total scale symptom score was lower than baseline
Progression-free survival (PFS) | 24 weeks
  PFS was defined as the time from date of randomization to disease progression radiological or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of disease evaluation.
Leukemia-free survival（LFS） | 24 weeks
  The time elapsed between the dates of any of the following events from a randomized solstice；The first bone marrow smear showed that the original cells were more than 20% of the date；The initial peripheral blood smear showed that the original cells were more than 20% and A peripheral blood blast content of 20% associated with an absolute blast count of 1*10(9)/L that lasts for at least 2 weeks；Death from any cause. Subjects without anyone of events at the time of analysis were censored at their last date of disease evaluation.
Overall survival (OS) | 2 years
  OS is defined as the time from date of randomization to death due to any cause. Subjects without death at the time of analysis were censored at their last date of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, MD, Study Chair — The First Affiliated Hospital of Medical School of Zhejiang University
Locations (1):
- The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share date of the trial